CLINICAL TRIAL: NCT04985318
Title: Retrospective Analysis of the Efficiency of Caplacizumab in the Treatment of Acquired Thrombotic Thrombocytopenic Purpura (aTTP)- REACT-2020
Brief Title: Retrospective Analysis of the Efficiency of Caplacizumab in the Treatment of aTTP
Acronym: REACT-2020
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Paul Brinkkoetter, Prof. MD, Consultant in Nephrology, University of Cologne
Other Study IDs: V01-19052020
Record Dates: First submitted 2021-07-21; First posted 2021-08-02 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acquired Thrombotic Thrombocytopenic Purpura
Keywords: aTTP; caplacizumab
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — caplacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registergroup: Patients with acquired Thrombotic Thrombocytopenic Purpura, who have been treated with caplacizumab (Cablivi®)
  Interventions: Drug: Cablivi®

INTERVENTIONS:
Drug: Cablivi® — Intervention with Cablivi® take place outside of the study

SUMMARY:
The objective of this national, prospective, multi-centre observational study is to describe the prescription rational and practice in Germany, confirm the efficacy of caplacizumab in a real-world setting, and identify predicting factors in iTTP-patients with regard to persistent autoimmune activity, therapy guidance and risk of complications. The rational is to develop new treatment algorithms that optimize overall patient outcome and reduce treatment cost.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of an acute episode of acquired thrombotic thrombocytopenic purpura
* Treatment with at least one single dose of caplacizumab (10 mg i.v. or s.c.)
* Male or female patients ≥ 18 years of age
* signed written informed consent

Exclusion Criteria:

* Hereditary thrombotic thrombocytopenic purpura
* disability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female subjects with confirmed diagnosis of an acute episode of aquired thrombotic thrombocytopenic purpura, who have been treated with one dose of caplacizumab.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2034-12-12 (Estimated); Study Completion 2034-12-12 (Estimated)

PRIMARY OUTCOMES:
Treatment of aTTP with caplacizumab | Enrollment
  Description of the prescription rationale and practice of caplacizumab in the treatment of aTTP

SECONDARY OUTCOMES:
Stabilization of thrombocyte | Enrollment
  Documentation of the efficacy of caplacizumab in the treatment of aTTP outside of clinical trials (real-world data) using by means of stabilization of thrombocyte. Thrombocyte stabilization is defined as thrombocyte > 150 x 10E9/L
Normalization of LDH | Enrollment
  Documentation of the efficacy of caplacizumab in the treatment of aTTP outside of clinical trials (real-world data) using by means of normalization of Lactate dehydrogenase (LDH). Normalization of LDH is defined as LDH below upper limit of normal
Normalization of haptoglobin | Enrollment
  Documentation of the efficacy of caplacizumab in the treatment of aTTP outside of clinical trials (real-world data) using by means of normalization of haptoglobin. Normalization of haptoglobin is defined as haptoglobin above lower limit of normal
Risk factors for complications | Enrollment
  Identification of risk factors for complications
Risk factors for adverse outcomes | Enrollment
  Identification of risk factors for adverse outcomes
Risk factors for persistent autoimmune activity | Enrollment
  Identification of risk factors for persistent autoimmune activity
Parameters for therapy guidance | Enrollment
  Identification of parameters that guide duration and regimen of caplacizumab treatment
Effect of caplacizumab on adjunct treatments with PEX | Enrollment
  Descriptions of the effect of caplacizumab on dose, duration and number and severity of adverse events of therapeutic plasma exchange therapy (PEX)
Effect of caplacizumab on adjunct treatments | Enrollment
  Descriptions of the effect of caplacizumab on dose, duration and number and severity of adverse events of glucocorticoids

CONTACTS AND LOCATIONS:
Overall Officials: Linus Völker, MD, Principal Investigator — Department II of Internal Medicine, University of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Volker LA, Kaufeld J, Balduin G, Merkel L, Kuhne L, Eichenauer DA, Osterholt T, Hagele H, Kann M, Grundmann F, Kolbrink B, Schulte K, Gackler A, Kribben A, Boss K, Potthoff SA, Rump LC, Schmidt T, Muhlfeld AS, Schulmann K, Hermann M, Gaedeke J, Sauerland K, Bramstedt J, Hinkel UP, Miesbach W, Bauer F, Westhoff TH, Bruck H, Buxhofer-Ausch V, Muller TJ, Wendt R, Harth A, Schreiber A, Seelow E, Tolle M, Gohlisch C, Bieringer M, Geuther G, Jabs WJ, Fischereder M, von Bergwelt-Baildon A, Schonermarck U, Knoebl P, Menne J, Brinkkoetter PT; German TTP-Study Group. Impact of first-line use of caplacizumab on treatment outcomes in immune thrombotic thrombocytopenic purpura. J Thromb Haemost. 2023 Mar;21(3):559-572. doi: 10.1016/j.jtha.2022.11.010. Epub 2022 Dec 22. PMID 36696206